CLINICAL TRIAL: NCT04181632
Title: Evaluation of Pain Alleviating Strategies During Allergy Shots (Subcutaneous Immunotherapy): A Randomized Controlled Study (Pain Perception With Allergy Shot Techniques: PPAST)
Brief Title: Evaluation of Pain Alleviating Strategies During Allergy Shots
Acronym: PPAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Jennifer Pfieffer, Pediatric Clinical Nurse Specialist, APRN, and Nurse Manager, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1353562
Record Dates: First submitted 2019-05-24; First posted 2019-11-29 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Immunotherapy; Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Study Design and Duration This is a randomized controlled study. Approximately 100 children, age 4 - 17 years, who are currently receiving subcutaneous immunotherapy, will randomly select a blinded envelope which assigns the distraction technique to be utilized during their study participation. There will be 25 envelopes assigned to each study group for a total of 100 envelopes. Each envelope will contain a paper with a colored sticker for the associated group assignment and number sequence.
  The distribution of group assignment by number sequence and color is as follows:
  Interventional Groups
  1. Shot Blocker® Number 1-25 (RED)
  2. Buzzy I® (vibrating only) Number 26-50 (GREEN)
  3. Buzzy II® (vibrating and ice wings) Number 51-75 (BLUE)
  4. Control Group Ethyl Chloride/Pain Ease Spray Number 76-100 (YELLOW)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Shot Blocker (Active Comparator): The three interventional groups are currently marketed distraction devices. Arm 1 will be Shot Blocker® Number 1-25 (RED).
  Interventions: Device: Shot Blocker
- Control Group (No Intervention): The control group is the current clinical standard of care option for pre-allergy injection application. Ethyl Chloride/Pain Ease Spray Number 76-100 (YELLOW).
- Buzzy I (Active Comparator): The three interventional groups are currently marketed distraction devices. Arm 2 will be Buzzy® I (vibrating only) Number 26-50 (GREEN).
  Interventions: Device: Buzzy Bee without Ice pack
- Buzzy II (Active Comparator): The three interventional groups are currently marketed distraction devices. Arm 3 will be Buzzy® II (vibrating and ice wings) Number 51-75 (BLUE).
  Interventions: Device: Buzzy Bee with Ice pack

INTERVENTIONS:
Device: Buzzy Bee with Ice pack — Buzzy uses natural pain relief to block needle pain for blood draws and shots. This intervention will be used with an ice pack.
  Arms: Buzzy II
Device: Buzzy Bee without Ice pack — Buzzy uses natural pain relief to block needle pain for blood draws and shots. This intervention will be used without an ice pack.
  Arms: Buzzy I
Device: Shot Blocker — Shot Blocker is a device that instantly alleviates the pain and anxiety of needle injections when pressed firmly against the skin at the injection site.
  Arms: Shot Blocker

SUMMARY:
Subcutaneous Immunotherapy (allergy injections) is a potentially disease-modifying therapy that is effective for the treatment of allergic rhinitis/conjunctivitis, allergic asthma and stinging insect hypersensitivity. Pain, which results from the irritation of nearby nerves is a common concern of patients, particularly in children, during or after the injections. This can be a stressful and negative experience for the children. There are various techniques available to minimize pain in general. However, there is a lack of published research on how to use these techniques in children receiving allergy injections. The purpose of this study is to evaluate and compare the efficacy of the standard of care method (Ethyl Chloride/Pain Ease Spray) and three non-pharmacological pain control devices (Buzzy Bee® I, Buzzy Bee II and Shot Blocke®r) in decreasing the perception of pain during subcutaneous allergy injection in a pediatric allergy/immunology clinic setting.

DETAILED DESCRIPTION:
This is a randomized controlled study. Approximately 100 children, age 4 - 17 years, who are currently receiving subcutaneous immunotherapy, will randomly select a blinded envelope which assigns the distraction technique to be utilized during their study participation. There will be 25 envelopes assigned to each study group for a total of 100 envelopes. Each envelope will contain a paper with a colored sticker for the associated group assignment and number sequence.

The distribution of group assignment by number sequence and color is as follows:

Interventional Groups

1. Shot Blocker® Number 1-25 (RED)
2. Buzzy I® (vibrating only) Number 26-50 (GREEN)
3. Buzzy II® (vibrating and ice wings) Number 51-75 (BLUE) Control Group
4. Ethyl Chloride/Pain Ease Spray Number 76-100 (YELLOW)

The three interventional groups are currently marketed distraction devices. The control group is the current clinical standard of care option for pre-allergy injection application.

The study consists of two visits. Both visits will be conducted during the participants routine clinic visit for allergy injections. At the first visit the investigator will assess eligibility. An overview of the study requirements will be provided to parent/child and consent/assent will be obtained.

During the second visit, the child will be randomized to a distraction technique or standard of care group to be utilized with the allergy injection(s) administered at this visit. Adherence with institutional allergy injection guidelines will be maintained. Prior to the application of the distraction method, the investigator will interview the parent to collect data related to demographic information and their child's current allergy health and treatment regime. The child's pain perception will be assessed before and after the allergy injection. The parent's perception of their child's pain will be assessed after the allergy injection. The investigator will provide information on the application of the randomized method and will provide instruction on the completion of the pain scales and questionnaires. The investigator and study staff will not indicate a method preference or guide the child or parent with their pain level responses. After completion of the second visit, the child's study participation is complete.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-17 years on injection immunotherapy
* A minimum of three allergy injection injections prior to enrollment at Visit 1
* Child accompanied by parent or legal guardian

Exclusion Criteria:

* Children with a known pain or sensory disorders
* Developmental delays lacking necessary cognitive ability
* Administration of any form of pain analgesic within eight hours of randomization at Visit 2

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Goal was to recruit 100 for sample size; however with COVID - only 40 were enrolled.
Period: Overall Study
Arm/Group | Shot Blocker | Control Group | Buzzy I | Buzzy II
Started | 12 | 9 | 8 | 11
Completed | 12 | 9 | 8 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shot Blocker | Control Group | Buzzy I | Buzzy II | Total
Number analyzed (Participants) | 12 | 9 | 8 | 11 | 40
Age, Customized [Median (Full Range); unit: years]
  Age Range | 14 [4 to 17] | 14 [4 to 17] | 12 [4 to 17] | 13 [4 to 17] | 13 [4 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 5 | 8 | 22
  Male | 6 | 6 | 3 | 3 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 5 | 4 | 7 | 22
  Black | 3 | 2 | 2 | 0 | 7
  Hispanic | 2 | 1 | 2 | 1 | 6
  Mixed/Other | 1 | 1 | 0 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 8 | 11 | 40
Pain Perception Before Allergy Shot [Mean (Standard Deviation); unit: units on a scale] — The change in patient pain perception will be captured utilizing the Wong-Baker FACES (actual faces of happiness or sadness etc. on the scale) Pain Rating Scale (0 no pain - 10 most pain) with each distraction method. The lower score is the better outcome.
  units on a scale | 0 (0) | 0.22 (0.67) | 0.0 (0.0) | 0 (0) | 0.05 (0.32)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Pain Perception Utilizing Three Non-pharmacological Pain Control / Distraction Devices and Ethyl Chloride Spray
Description: The change in patient pain perception will be captured utilizing the Wong-Baker FACES (actual faces of happiness or sadness etc. on the scale) Pain Rating Scale (0 no pain - 10 most pain) with each distraction method. The lower score is the better outcome.
Time Frame: Assessment of pain perception before and within 1 minute after the application of the distraction method and administration of the allergy injection within their 30-minute allergy shot appointment.
Population: Results A total of 40 children who received SCIT were included in this randomized controlled pilot study. Of these 40 children, 12 received the ShotBlocker, 8 received the Buzzy I, 11 received the Buzzy II, and 9 received ethyl chloride spray (control group). Both the overall needle pain rating by the children after their allergy injection and the overall parental perception of needle pain are displayed by each of the four interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shot Blocker | Control Group | Buzzy I | Buzzy II
Number analyzed (Participants) | 12 | 9 | 8 | 11
score on a scale | 1.33 (1.3) | 2.22 (2.11) | 2.25 (1.28) | 1.45 (1.57)

ADVERSE EVENTS:
Time Frame: 30 minutes
Arm/Group | Shot Blocker | Control Group | Buzzy I | Buzzy II
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/8 | 0/11

LIMITATIONS AND CAVEATS:
COVID, decreased enrollment, clinic closed, etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT04181632/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT04181632/ICF_001.pdf